CLINICAL TRIAL: NCT03998566
Title: Early Feasibility Study For Evaluation Of The TraceIT® Tissue Spacer For Creating Space Between The Duodenum And Pancreas In Patients With Localized Pancreatic Cancer Undergoing Radiation Therapy
Brief Title: Radiopaque Hydrogel Spacer in Patients Undergoing Radiotherapy for Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGX17-001-US
Record Dates: First submitted 2019-06-13; First posted 2019-06-26 (Actual); Results first posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Pancreatic Cancer
Keywords: Radiotherapy; Radiation; SBRT
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- TraceIT Tissue Spacer (Experimental)
  Interventions: Device: TraceIT Tissue Spacer implantation

INTERVENTIONS:
Device: TraceIT Tissue Spacer implantation — The TraceIT Tissue Spacer will be implanted between duodenum and pancreas using endoscopic procedure. After implantation patient will have radiotherapy treatment per standard of care.

SUMMARY:
An early feasibility study to evaluate feasibility, radiotherapy benefits and safety when using TraceIT tissue spacer to create space between pancreas and duodenum in patients with localized Pancreatic Cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Biopsy-confirmed localized pancreatic cancer in the head or neck of the pancreas as defined by the NCCN guidelines
3. Tumor is clearly delineable from duodenum and no clear evidence of invasion of the duodenum is seen at time of EUS performed for either diagnosis or fiducial placement.
4. Subject is able to comply with motion management guidelines.
5. Radiotherapy or chemoradiotherapy for treatment of the disease is indicated.
6. In Investigator's opinion, medically fit to undergo endoscopy for fiducial marker implantation and TraceIT administration.
7. Subjects Screening/Baseline laboratory testing must meet the following laboratory value criteria:

   1. White blood cell count: ≥ 3.0 x 109/L
   2. Absolute neutrophil count (ANC): ≥ 1.5 x 109/L
   3. Platelets: ≥ 100 x 109/L
   4. Total bilirubin: ≤ 2.0 times upper limit of normal (ULN)
   5. AST and ALT: ≤ 3.0 times institutional upper normal limit
   6. Serum creatinine: < 1.5 times ULN e
   7. INR: < 1.5
   8. Serum pregnancy: Negative
   9. Hemoglobin: ≥ 8.0 g/dl
8. Zubrod Performance Status 0-2
9. Subject or authorized representative, has been informed of the nature of the study and has provided written informed consent, approved by the appropriate Institutional Review Board (IRB) of the respective clinical site.
10. Life expectancy of at least 9 months

Exclusion Criteria:

1. Patients for whom radiotherapy is contraindicated
2. Previous thoracic or abdominal radiotherapy
3. Any GI abnormality that would interfere with the ability to access the injection site
4. Presence of tumor invasion of the duodenum detected on EUS at time of biopsy
5. Previous Whipple procedure or other resection of pancreatic tumor prior to screening
6. Active gastroduodenal ulcer or uncontrolled watery diarrhea
7. History of Chronic Renal Failure.
8. Documented history of uncontrolled diabetes (i.e., symptomatic hyperglycemia that cannot be medically managed, fasting blood glucose level above 300 mg/dL, and/or frequent swings between hyperglycemia and hypoglycemia)
9. Currently enrolled in another investigational drug or device trial that clinically interferes with this study.
10. Unable to comply with the study requirements or follow-up schedule.
11. Any condition or comorbidity that the Investigator believes would interfere with the intent of the study or would make participation not in the best interest of the subject.
12. Women who are pregnant or breast-feeding; women of child-bearing age must use contraceptives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Johns Hopkins Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TraceIT Tissue Spacer
Started | 6
Completed | 1
Not Completed | 5

BASELINE CHARACTERISTICS:
Population: Modified Intent to Treat (MITT)
Arm/Group | TraceIT Tissue Spacer
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Safety Endpoint
Description: Number of subjects with TraceIT procedure-related event which resulted in a delay in initiation for RT (radio-therapy).
Time Frame: 2-6 week assessment post-procedure
Population: Modified Intent to Treat (MITT)
Measure: Count of Participants; unit: Participants
Groups:
- All TIPS Participant: Subjects with localized (resectable, borderline resectable or locally advanced) pancreatic cancer (defined per NCCN guidelines) that have completed induction chemotherapy if required and for whom a course of radiotherapy (RT) was indicated.
Arm/Group | All TIPS Participant
Number analyzed (Participants) | 6
Participants
  No | 6
  Yes | 0

2. Secondary Outcome: Radio-Therapy Benefits of TraceIT
Description: Number of subjects who were able to maintain safe duodenal dose constraints. RT benefits were assessed via comparison of pre- and post-TraceIT administration RT plans with consideration of the following: ability to maintain safe duodenal dose constraints, percent/volume of gross tumor volume/planning target volume (GTV/PTV) receiving prescription dose and overall duodenal dose/dose distribution.
Time Frame: 2-6 week assessment
Population: Modified Intent to Treat (MITT)
Measure: Count of Participants; unit: Participants
Groups:
- All TIPS Participants: Subjects with localized (resectable, borderline resectable or locally advanced) pancreatic cancer (defined per NCCN guidelines) that have completed induction chemotherapy if required and for whom a course of radiotherapy (RT) was indicated.
Arm/Group | All TIPS Participants
Number analyzed (Participants) | 6
Participants
  Yes | 6
  No | 0

3. Secondary Outcome: Feasibility of TraceIT
Description: Number of subjects who achieved Technical Success (the ability to place TraceIT and create space between the duodenum and head of pancreas (HOP).
Time Frame: 2-6 week assessment post-procedure
Population: Modified Intent to Treat (MITT)
Measure: Count of Participants; unit: Participants
Arm/Group | All TIPS Participant
Number analyzed (Participants) | 6
Participants
  Yes | 6
  No | 0

4. Secondary Outcome: TraceIT Persistence (at 6-months Post-treatment)
Description: Characteristics of TraceIT persistence and migration were measured at 2 to 6 weeks and 6 months following injection. Persistence was measured at the 2 to 6 week and 6 month follow-ups by assessing whether a cohesive mass of water density fluid was present in the periduodenal space following the last radio therapy appointment. Migration of the TraceIT post Radiation was measured by CT scan taken at 2-6 weeks follow-up.
Time Frame: 2-6 weeks and 6 month post procedure
Population: Modified Intent to Treat (MITT)
Measure: Count of Participants; unit: Participants
Groups:
- 2-3 Weeks Follow-up Post Radiation Therapy; 6 Month Follow-up Post Radiation Therapy: Number of subjects showing persistence and migration.
Arm/Group | 2-3 Weeks Follow-up Post Radiation Therapy | 6 Month Follow-up Post Radiation Therapy
Number analyzed (Participants) | 6 | 6
Participants
  Persistence: number analyzed (Participants) | 3 | 2
  Persistence: No | 0 | 2
  Persistence: Yes | 3 | 0
  Migration: number analyzed (Participants) | 5 | 0
  Migration: No | 3 |
  Migration: Yes | 2 |

5. Secondary Outcome: Theoretical Dose Escalation From Post-TraceIT Treatment Plan
Description: Maximum dose to the GTV while maintaining duodenal dose constraints
Time Frame: 2-6 week assessment Post-procedure
Population: Modified Intent to Treat (MITT)
Measure: Mean (Standard Deviation); unit: Gy
Arm/Group | All TIPS Participants
Number analyzed (Participants) | 6
Gy | 12.7 (19.7)

6. Secondary Outcome: Incidence of Acute (Within 3 Months) and Late (>3 Months) Duodenal Toxicity Summarized by CTCAE Grade and Timing
Description: Number of subject with Duodenal AE summarized by CTCAE grade and timing
Time Frame: 18 months post procedure
Population: Modified Intent to Treat (MITT)
Measure: Number; unit: participants
Groups:
- Total: Total number of subjects
- One or More Acute (<=3 Months): Subjects who have experienced one or more acute AEs within 3 months of index procedure.
- One or More Late (>3 Months): Subjects who have experienced one or more AEs more than 3 months after index procedure.
Arm/Group | Total | One or More Acute (<=3 Months) | One or More Late (>3 Months)
Number analyzed (Participants) | 6 | 6 | 6
participants
  Subjects who have one or more grade 1 duodenal AEs | 6 | 6 | 4
  Subjects who have one or more grade 2 duodenal AEs | 4 | 3 | 3
  Subjects who have one or more grade 3 duodenal AEs | 2 | 0 | 2
  Subjects who have one or more grade 4 duodenal AEs | 0 | 0 | 0
  Subjects who have one or more grade 5 duodenal AEs | 0 | 0 | 0
  Subjects who only have grade N/A duodenal AEs | 0 | 0 | 0
  Subjects who have one or more duodenal AEs | 6 | 6 | 4

7. Secondary Outcome: Incidence of Resection Following the Completion of Radiation Therapy (RT)
Description: Number of subjects with resection following the completion of radiation therapy (RT). Within 2-6 weeks after completion of therapy, subjects were restaged to determine whether they may progress for surgery (resection).
Time Frame: 2-6 weeks post procedure
Population: Modified Intent to Treat (MITT)
Measure: Count of Participants; unit: Participants
Arm/Group | All TIPS Participants
Number analyzed (Participants) | 6
Participants
  Yes | 3
  No | 3

8. Secondary Outcome: Progression Free and Overall Survival
Description: Progression-free survival is the interval between the start of induction chemotherapy (prior to Radiation Therapy) to the earliest treatment failure onset date, or death, in months. Overall survival is the interval between the start of induction chemotherapy (prior to radiation therapy) to death in month.
Time Frame: 18 months post procedure
Population: Modified Intent to Treat (MITT)
Measure: Mean (Standard Deviation); unit: months
Arm/Group | All TIPS Participants
Number analyzed (Participants) | 6
months
  Progression free survival (subjects with tumor progression event): number analyzed (Participants) | 3
  Progression free survival (subjects with tumor progression event) | 17.6 (4.7)
  Overall survival in subjects who died: number analyzed (Participants) | 3
  Overall survival in subjects who died | 20.0 (10.1)

9. Secondary Outcome: Changes From Baseline at the Final RT Appointment, 3 Month, 6 Month, 12 Month and 18 Month in EORTC QoL (QLQ-C30)
Description: The EORTC QOL QLQ-C30 is a questionnaire used to assess patient-reported symptoms and outcomes during cancer treatment. The survey contains 28 questions scored on a 4-point Likert scale (1 = 'Not at all' to 4 'Very much') and 2 questions on a 7-point numerical scale (1 = 'Very poor' to 7 = 'Excellent').Questions are grouped into 15 categories containing 1 to 5 different questions per category. All scores were transformed to a 0-100 scale following instructions in the scoring manual. Raw scores calculated as the average of component items are then standardized using linear transformation to a score ranging from 0-100. Higher score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/QoL represents a high QoL. A high score for a symptom scale/item represents a high level of symptomatology/problems.
Time Frame: Changes in baseline at the Final RT appointment, 3 month, 6 month, 12 month and 18 month
Population: Modified Intent to Treat (MITT)
Measure: Mean (Full Range); unit: Scores on a scale
Groups:
- Final RT: Subjects with localized (resectable, borderline resectable or locally advanced) pancreatic cancer (defined per NCCN guidelines) that have completed induction chemotherapy if required and for whom a course of radiotherapy (RT) was indicated.
- 3 Months: Subject outcomes at 3 month follow-up visit
- 6 Month: Subject outcome at 6 month follow-up visit
- 12 Month: Subject outcomes at 12 Month follow-up visit
- 18 Month: Subject outcome at 18 month follow-up visit
Arm/Group | Final RT | 3 Months | 6 Month | 12 Month | 18 Month
Number analyzed (Participants) | 6 | 6 | 6 | 4 | 1
Scores on a scale
  Change of Global health status: number analyzed (Participants) | 5 | 3 | 5 | 2 | 1
  Change of Global health status | -6.7 [-25 to 0] | -11.1 [-25 to 8.3] | 3.3 [-33.3 to 25] | -29.2 [-33.3 to -25] | 0 [0 to 0]
  Physical functioning: number analyzed (Participants) | 5 | 3 | 5 | 2 | 1
  Physical functioning | 1.3 [0 to 6.7] | -17.8 [-46.7 to 0] | 1.3 [-13.3 to 20] | -10.0 [-20 to 0] | -13.3 [-13.3 to -13.3]
  Role Functioning: number analyzed (Participants) | 5 | 3 | 5 | 2 | 1
  Role Functioning | -13.3 [-33.3 to 0] | -50.0 [-100 to 0] | 0 [-33.3 to 0] | -8.3 [-16.7 to 0] | -66.7 [-66.7 to -66.7]
  Emotional Functioning: number analyzed (Participants) | 5 | 3 | 5 | 2 | 1
  Emotional Functioning | -5 [-33.3 to 8.3] | 5.6 [0 to 8.3] | 6.7 [-25 to 25] | -20.8 [-25 to -16.7] | -33.3 [-33.3 to -33.3]
  Cognitive Functioning: number analyzed (Participants) | 5 | 3 | 5 | 2 | 1
  Cognitive Functioning | 0 [-16.7 to 33.3] | -16.7 [-50 to 0] | 3.3 [0 to 16.7] | -8.3 [-16.7 to 0] | -33.3 [-33.3 to -33.3]
  Social Functioning: number analyzed (Participants) | 5 | 3 | 5 | 2 | 1
  Social Functioning | 20 [0 to 50] | -5.6 [-16.7 to 0] | 16.7 [-16.7 to 50] | -16.7 [-33.3 to 0] | -66.7 [-66.7 to -66.7]
  Fatigue: number analyzed (Participants) | 5 | 3 | 5 | 2 | 1
  Fatigue | 11.1 [0 to 33.3] | 37 [0 to 66.7] | 11.1 [0 to 33.3] | 0 [0 to 0] | 33.3 [33.3 to 33.3]
  Nausea and Vomiting: number analyzed (Participants) | 5 | 3 | 5 | 2 | 1
  Nausea and Vomiting | 13.3 [0 to 33.3] | 5.6 [0 to 16.7] | -6.7 [-16.7 to 0] | 0 [0 to 0] | 16.7 [16.7 to 16.7]
  Pain: number analyzed (Participants) | 5 | 3 | 5 | 2 | 1
  Pain | 3.3 [-16.7 to 16.7] | 0 [0 to 0] | -10 [-16.7 to 0] | -8.3 [-16.7 to 0] | 50 [50 to 50]
  Dyspnea: number analyzed (Participants) | 5 | 3 | 5 | 2 | 1
  Dyspnea | -13.3 [-33.3 to 0] | -11.1 [-33.3 to 0] | -20 [-66.7 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Insomnia: number analyzed (Participants) | 5 | 3 | 5 | 2 | 1
  Insomnia | -6.7 [-66.7 to 33.3] | 11.1 [0 to 33.3] | 0 [-33.3 to 33.3] | 16.7 [0 to 33.3] | 33.3 [33.3 to 33.3]
  Appetite loss: number analyzed (Participants) | 5 | 3 | 5 | 2 | 1
  Appetite loss | 6.7 [-33.3 to 33.3] | 33.3 [0 to 66.7] | 6.7 [0 to 33.3] | 0 [0 to 0] | 66.7 [66.7 to 66.7]
  Constipation: number analyzed (Participants) | 5 | 3 | 5 | 2 | 1
  Constipation | 13.3 [0 to 66.7] | -22.2 [-33.3 to 0] | -13.3 [-33.3 to 0] | 0 [0 to 0] | 33.3 [33.3 to 33.3]
  Diarrhea: number analyzed (Participants) | 5 | 3 | 5 | 1 | 1
  Diarrhea | 6.7 [0 to 33.3] | 0 [-33.3 to 33.3] | -6.7 [-33.3 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Financial Difficulties: number analyzed (Participants) | 5 | 3 | 5 | 2 | 1
  Financial Difficulties | 6.7 [0 to 33.3] | -11.1 [-33.3 to 0] | 0 [-33.3 to 33.3] | 16.7 [0 to 33.3] | 0 [0 to 0]

10. Other Pre Specified Outcome: Comparability of Visualization of the Fiducial Marker and TraceIT Hydrogel
Description: Scores for the visualization of the fiducial marker and TraceIT hydrogel.
Time Frame: 2-5 weeks assessment post procedure
Population: Modified Intent to Treat (MITT)
Measure: Count of Participants; unit: Participants
Arm/Group | All TIPS Participants
Number analyzed (Participants) | 6
Participants
  Fiducial marker visibility scoring: 1-Not visualized | 0
  Fiducial marker visibility scoring: 2-Faint or trace visibility (shadow or haze) | 0
  Fiducial marker visibility scoring: 3-Visibility but indistinct borders (definable entity) | 0
  Fiducial marker visibility scoring: 4-Partially distinct border, partial haze | 1
  Fiducial marker visibility scoring: 5- Clearly visualized, unequivocal | 5
  TraceIT hydrogel visibility scoring: 1-Not visualized | 0
  TraceIT hydrogel visibility scoring: 2-Faint or trace visibility (shadow or haze) | 0
  TraceIT hydrogel visibility scoring: 3-Visibility but indistinct borders (definable entity) | 2
  TraceIT hydrogel visibility scoring: 4-Partially distinct border, partial haze | 0
  TraceIT hydrogel visibility scoring: 5- Clearly visualized, unequivocal | 4

11. Other Pre Specified Outcome: TraceIT Stability and Space Measurements
Description: The stability of TraceIT was measured as the minimum distance from the fiducial marker to TraceIT gel. Space measurements were taken before and after TraceIT was injected, which measured the preduodenal space using the axial view along the head of the HOP.
Time Frame: Pre-TraceIT and Post-TraceIT procedure, up to 2-6 weeks follow-up post radiation therapy
Population: Modified Intent to Treat (MITT)
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Pre-TraceIT: Space measurements taken before TraceIT was injected.
- Post- TraceIT: Stability measured as the minimum distance from the fiducial maker to TraceIT gel.
  Space measurement taken after TraceIT was injected.
- 2-6 Weeks Follow-up Post Radiation Therapy: Stability measured as the minimum distance from the fiducial maker to TraceIT gel.
Arm/Group | Pre-TraceIT | Post- TraceIT | 2-6 Weeks Follow-up Post Radiation Therapy
Number analyzed (Participants) | 6 | 3 | 3
mm
  Stability - Minimum distance from fiducial to TraceIT gel (mm): number analyzed (Participants) | 0 | 3 | 3
  Stability - Minimum distance from fiducial to TraceIT gel (mm) |  | 8.2 (5.9) | 8.5 (10.2)
  TraceIT Space Measurement (mm): number analyzed (Participants) | 6 | 3 | 0
  TraceIT Space Measurement (mm) | 1.0 (0) | 7.7 (2.4) |

12. Other Pre Specified Outcome: Changes From Baseline Final RT Appointment, 3 Months, 6 Months, 12 Months, and 18 Months in QLQ-PAN26
Description: The QLQ-PAN26 questionnaire is a survey designed to assess patient-reported symptoms of patients undergoing treatment for pancreatic cancer. All of the scales and single item measures range in score from 0-100. A high score for the symptom scales and/or single items represents a high level of symptomatology or problems, whereas a high score for the functional scales represents a high level of functioning.
Time Frame: Changes from baseline final RT appointment, 3 months, 6 months, 12 months, and 18 months in QLQ-PAN26
Population: Modified Intent to Treat
Measure: Mean (Full Range); unit: score on a scale
Groups:
- 18 Month: Subject outcome 18 month follow-up visit
Arm/Group | Final RT | 3 Months | 6 Month | 12 Month | 18 Month
Number analyzed (Participants) | 6 | 6 | 6 | 4 | 1
score on a scale
  Pancreatic Pain: number analyzed (Participants) | 5 | 3 | 5 | 1 | 1
  Pancreatic Pain | 1.7 [-8.3 to 25] | 2.8 [0 to 8.3] | -10 [-25 to 0] | 8.3 [8.3 to 8.3] | 8.3 [8.3 to 8.3]
  Bloating: number analyzed (Participants) | 5 | 3 | 5 | 1 | 1
  Bloating | 0 [-33.3 to 33.3] | 11.1 [0 to 33.3] | -6.7 [-33.3 to 0] | 33.3 [33.3 to 33.3] | 0 [0 to 0]
  Digestive Symptoms: number analyzed (Participants) | 5 | 3 | 5 | 1 | 1
  Digestive Symptoms | 30 [0 to 50] | 44.4 [0 to 100] | 26.7 [0 to 66.7] | -16.7 [-16.7 to -16.7] | 66.7 [66.7 to 66.7]
  Taste: number analyzed (Participants) | 5 | 3 | 5 | 1 | 1
  Taste | 6.7 [0 to 33.3] | 66.7 [33.3 to 100] | -6.7 [-33.3 to 66.7] | -33.3 [-33.3 to -33.3] | 33.3 [33.3 to 33.3]
  Indigestion: number analyzed (Participants) | 5 | 3 | 5 | 1 | 1
  Indigestion | 0 [0 to 0] | 0 [0 to 0] | -26.7 [-66.7 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Flatulence: number analyzed (Participants) | 5 | 3 | 5 | 1 | 1
  Flatulence | 33.3 [0 to 66.7] | 0 [-33.3 to 33.3] | 13.3 [-33.3 to 66.7] | 0 [0 to 0] | 0 [0 to 0]
  Weight Loss: number analyzed (Participants) | 5 | 3 | 5 | 1 | 1
  Weight Loss | 0 [0 to 0] | 11.1 [0 to 33.3] | 0 [0 to 0] | 33.3 [33.3 to 33.3] | 33.3 [33.3 to 33.3]
  Weakness arms and legs: number analyzed (Participants) | 5 | 3 | 5 | 1 | 1
  Weakness arms and legs | 0 [-33.3 to 33.3] | 22.2 [0 to 33.3] | 13.3 [0 to 33.3] | 33.3 [33.3 to 33.3] | 33.3 [33.3 to 33.3]
  Dry Mouth: number analyzed (Participants) | 5 | 3 | 5 | 1 | 1
  Dry Mouth | -6.7 [-33.3 to 0] | 22.2 [-33.3 to 100] | -13.3 [-33.3 to 0] | 33.3 [33.3 to 33.3] | -33.3 [-33.3 to -33.3]
  Hepatic Symptoms: number analyzed (Participants) | 5 | 3 | 5 | 1 | 1
  Hepatic Symptoms | -10 [-33.3 to 0] | -5.6 [-16.7 to 0] | -3.3 [-16.7 to 0] | 50 [50 to 50] | -16.7 [-16.7 to -16.7]
  Altered Bowel Habit: number analyzed (Participants) | 5 | 3 | 5 | 1 | 1
  Altered Bowel Habit | -3.3 [-83.3 to 66.7] | 22.2 [0 to 50] | -3.3 [-33.3 to 16.7] | 33.3 [33.3 to 33.3] | 16.7 [16.7 to 16.7]
  Body Image: number analyzed (Participants) | 5 | 3 | 5 | 1 | 1
  Body Image | 0 [-50 to 16.7] | -11.1 [-33.3 to 16.7] | 6.7 [-50 to 83.3] | 0 [0 to 0] | 50 [50 to 50]
  Trouble with side-effects: number analyzed (Participants) | 5 | 3 | 5 | 1 | 1
  Trouble with side-effects | -20 [-66.7 to 33.3] | 22.2 [0 to 66.7] | -6.7 [-33.3 to 33.3] | 66.7 [66.7 to 66.7] | 33.3 [33.3 to 33.3]
  Future Worries: number analyzed (Participants) | 5 | 3 | 5 | 1 | 1
  Future Worries | 20 [0 to 66.7] | -11.1 [-33.3 to 0] | 0 [-33.3 to 33.3] | 66.7 [66.7 to 66.7] | 33.3 [33.3 to 33.3]
  Planning of activities: number analyzed (Participants) | 5 | 3 | 5 | 1 | 1
  Planning of activities | -13.3 [-100 to 33.3] | 44.4 [0 to 100] | 20 [-33.3 to 66.7] | 0 [0 to 0] | 33.3 [33.3 to 33.3]
  Satisfaction with health care: number analyzed (Participants) | 5 | 3 | 5 | 1 | 1
  Satisfaction with health care | 6.7 [-33.3 to 50] | -5.6 [-16.7 to 0] | 10 [0 to 33.3] | 0 [0 to 0] | -16.7 [-16.7 to -16.7]
  Sexuality: number analyzed (Participants) | 5 | 3 | 5 | 1 | 1
  Sexuality | 0 [-33.3 to 33.3] | 0 [-33.3 to 33.3] | 0 [-33.3 to 50] | -33.3 [-33.3 to -33.3] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from initiation of fiducial marker placement through the 18 month visit.
Description: Adverse Events(AE), Adverse Device Effect (ADE),Serious Adverse Event (SAE), Serious Adverse Device Effect (SADE), and Unanticipated Adverse Device Effect (UADE) were collected.
  All AEs and SAEs,will be collected from the time of fiducial maker placement and through the 18-month visit. Subjects who experience an AE/SAEs related to TraceIT hydrogel will be followed until the AE has resolved or until the subject has stabilized and FU care has been transferred to subject's primary care physician.
Arm/Group | TraceIT Tissue Spacer
All-Cause Mortality (participants affected / at risk) | 3/6
Serious Adverse Events (participants affected / at risk) | 6/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TraceIT Tissue Spacer (N=6)
Abdominal Pain (Gastrointestinal disorders) | 3 (6)
Acute Cholangitis (Hepatobiliary disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Bile Duct Stenosis (Hepatobiliary disorders) | 1 (1)
Death due to Disease progression/worsening of Pancreatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Disease recurrence in the pancreas and metastasis to the lower lobe of the right lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Gastrointestinal disorder- Other (Gastrointestinal disorders) | 1 (1) — Cholangitis
Gastrointestinal disorders- Other (Gastrointestinal disorders) | 1 (1) — Obstructive hyperbilirubinemia
Gastrointestinal disorders- Other (Gastrointestinal disorders) | 1 (1) — Liver Abscess
Headache (Nervous system disorders) | 1 (1)
Hemorrhagic Stroke (Nervous system disorders) | 1 (1)
High Fever (General disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Infections and infestations- Other (Infections and infestations) | 1 (1) — bacterial peritonitis
Infections and infestations- Other (Infections and infestations) | 1 (1) — Influenza B
Infections and infestations- Other (Infections and infestations) | 1 (1) — Coronavirus HKU1
Investigations - Other, (Investigations) | 1 (1) — Blood Bilirubin Increased
Musculoskeletal and connective tissue disorder- Other (Musculoskeletal and connective tissue disorders) | 1 (1) — Right Thoracic Facet Spondylosis
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) — distant metastasis
Nervous system disorders- Other (Nervous system disorders) | 1 (1) — Cancer-Related Pain
Neuralgia (Nervous system disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (2)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Respiratory depression
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) — hypercapnic respiratory failure
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) — bacterial pneumonia
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) — pneumonia
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Surgical and medical procedures - Other (Surgical and medical procedures) | 1 (1) — Drain site erythema
Urinary tract infection (Infections and infestations) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TraceIT Tissue Spacer (N=6)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (10)
Alanine aminotransferase increased (Investigations) | 2 (4)
Alkaline phosphatase increased (Investigations) | 3 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 5 (9)
Anorexia (Metabolism and nutrition disorders) | 3 (5)
Anxiety (Psychiatric disorders) | 1 (1)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (4)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (1)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 (1) — Thrombocytopenia
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Cardiac disorders - Other (Cardiac disorders) | 1 (1) — pulmonary embolism
Chills (General disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Decreased Leukocytes - Grade 2 (Investigations) | 1 (1)
Decreased Neutrophils - Grade 2 (Investigations) | 1 (1)
Decreased Platelet Count - Grade 1 (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (4)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (8)
Disease Progression (General disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 2 (2)
Erythmatous Injection Sites (General disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Fatigue (General disorders) | 5 (9)
Fever (General disorders) | 4 (5)
Flatulence (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) — inguinal hernia
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) — Paraesophageal Hernia
General disorders and administration site conditions - Other (General disorders) | 1 (1) — Temperature regulation disorder
General disorders and administration site conditions - Other (General disorders) | 1 (1) — localized edema - lower extremity
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (5)
Hematoma (Vascular disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1 (1) — Hepatic steatosis
Hot flashes (Vascular disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2)
Hypertension (Vascular disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Ileus (Gastrointestinal disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Investigations - Other (Investigations) | 1 (1) — Blood bilirubin increased
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (7)
Malaise (General disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Mild Chest Cold (Infections and infestations) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) — Throracolumbar Spondylosis without Radiculopathy
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) — generalized muscle weakness
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) — abnormalities of gait
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) — decreased mobility
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) — left ankle pain
Nausea (Gastrointestinal disorders) | 5 (15)
Nervous system disorders - Other (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Occasional Leg Cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
Occasional Nausea (Gastrointestinal disorders) | 1 (1)
Occasional Vomiting (General disorders) | 1 (1)
Oral Thrush (Infections and infestations) | 1 (1)
Pain (General disorders) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain Near Incision Site (Injury, poisoning and procedural complications) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Platelet count decreased (Investigations) | 2 (3)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Pruiritic Injection Sites (General disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Psychiatric disorders - Other (Psychiatric disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2)
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 (1) — Glucosuria Present Grade 1
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 (1) — chronic renal insufficiency
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) — pneumonia
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) — reactive airway disease
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) — shortness of breath
Sinus bradycardia (Cardiac disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Vascular disorders - Other (Vascular disorders) | 1 (1) — swelling of leg (left)
Weight loss (Investigations) | 1 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/66/NCT03998566/Prot_003.pdf
  • Statistical Analysis Plan (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/66/NCT03998566/SAP_004.pdf